## CONSENT FORM A: RAS MUTATION STATUS and c-MET MUTATION/EXPRESSION SCREENING

Short Title: MErCuRIC1: MEK and MET Inhibition in Colorectal Cancer

REC Reference: 14/SC/1010

| Patient Statement and Signature To be completed by the patient You must agree to points 1-10 to enter the study Please initial the boxes | | |
|---|---|---|
| 1. | I confirm that I have received verbal information and read and understand the information sheet dated DD MON YYYYY, Version Number for the RAS mutation status and c-MET mutation, amplification or over-expression screening for the above study. | Initials |
| 2. | I have had the opportunity to consider the information and ask questions, and I have had these answered satisfactorily. | |
| 3. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason and without my medical care or legal rights being affected. | |
| 4. | I understand that relevant sections of any of my medical notes and data collected during the study may be looked at by responsible individuals from the University of Oxford, from my treating hospital and the regulatory agency who authorised the trial, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | |
| 5. | I agree that my data may be transferred outside the European Economic Area to countries which may have a lower level of Data Protection. | |
| 6. | I agree to my GP being informed of my participation in the study. | |
| 7. | If I (or my partner) become pregnant while receiving trial medication, or within 6 months of taking the last trial medication, I agree to provide the information requested on the pregnancy and the outcome of the pregnancy. | |
| 8. | I agree to have a new biopsy of my cancer from an accessible site. | |
| 9. | I agree to the use of my tumour sample that is stored in the pathology laboratory for screening. | |
| 10. | I agree to take part in mutation status and c-MET mutation, amplification or over-<br>expression screening for the above study. | |
| Optional If you agree please <u>initial</u> t | | |
| 11. | I agree to donate any leftover biological sample material from the tumour samples I provide for further research purposes. I consider these samples a gift to the University of Oxford and I understand I will not gain any direct personal benefit from them. I give permission for my samples and trial information to be stored in a licenced tissue bank for use in any ethically approved medical research. I understand that this requires a copy of this consent form, which will identify me by name, to be sent to the tissue bank. | |

| Your signature confirms that you have had an opportunity to ask questions and that all of your questions have been answered. You will be given a signed and dated copy of this consent form to take away with you. | | |
|---|---|---|
| Name of<br>Patient<br>(print): | Patient signature: | Date<br>signed: |
| Investigator Statement and Signature To be completed by the person taking consent | | |
| I have discussed this clinical research study with the patient using a language that is understandable and appropriate. I believe that I have fully informed the participant of the nature of this study and the possible benefits and risks of taking part. I believe the participant has understood this explanation. | | |
| Name of person taking consent (Print): | Signature<br>of person<br>taking<br>consent | Date<br>signed: |

When completed: Original for Investigator Site File; a copy for participant; a copy to be kept in medical notes; a copy to OCTO; a copy to the licenced tissue bank.